CLINICAL TRIAL: NCT02289313
Title: Development of a Youth Healthy Living Program at the Rochester Alternative Learning Center
Brief Title: Development of a Youth Healthy Living Program With Underserved Adolescents at Rochester Alternative Learning Center
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Rochester Alternative Learning Center (Unknown)
Responsible Party: Principal Investigator, Seema Kumar, MD, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 14-004474
Record Dates: First submitted 2014-11-09; First posted 2014-11-13 (Estimated); Last update posted 2021-12-16 (Actual); Status verified 2021-12

CONDITIONS: Childhood Obesity
Keywords: obesity prevention; CBPR; high risk youth; school health
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Youth Healthy Living Program (Experimental): Youth attending the Rochester Alternative Learning Center (ALC) will be enrolled in a youth healthy living program at the ALC.
  Interventions: Behavioral: Healthy Youth Living Program

INTERVENTIONS:
Behavioral: Healthy Youth Living Program — Physical activity and healthy eating program at the Alternative Learning Center co-developed by students, school staff and academic partners.

SUMMARY:
Approximately one third of the children and adolescents in the United States are either overweight or obese. Childhood obesity disproportionately affects specific racial and ethnic groups and households with low socioeconomic status and low parental education. The Alternative Learning Center (ALC) within Rochester School District 535 provides viable educational options for students who are experiencing difficulty in regular educational systems. A greater proportion of students at ALC are minorities, qualify for free and reduced lunch and receive special education services. These children are likely to have unique barriers to physical activity and healthy eating.

Specific Aims:

Aim 1: Examine the association between BMI and ethnic/ socioeconomic variables and behaviors related to physical activity and eating in ALC students.

Aim 2: Develop an age and culturally appropriate on-site program that promotes healthy lifestyle.

DETAILED DESCRIPTION:
Investigators will assess the relationship between BMI and ethnicity, socioeconomic variables and behaviors related to nutrition and physical activity among 200 ALC students. Investigators will also conduct 6 gender stratified (3 boys, 3 girls) focus groups with students (n=24), up to 3 focus groups with their parents (n=24) and one focus group with staff and volunteers in order to understand perceived barriers towards healthy weight/nutrition/physical activity. Investigators will then utilize this information to co-develop a healthy living program at ALC. Investigators will finally test the feasibility of the program they develop over a period of 3 months in ALC students. Study findings will inform further research to test the efficacy and validity of the program developed at ALC in a subsequent school based trial with the future goal of obtaining funding for cluster randomized controlled trials among other schools in the region.

ELIGIBILITY:
Inclusion criteria:

* Rochester Alternative Learning Center students ages 12 years to 20 years
* Parents/guardians of ALC students
* ALC staff.

Exclusion criteria:

* Inability to assent or consent to participate in the study.

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2014-11; Primary Completion 2015-03-06 (Actual); Study Completion 2015-06-17 (Actual)

PRIMARY OUTCOMES:
Behaviors related to healthy eating and physical activity | 3 months
  Adoption of healthy eating choices by Rochester Alternative Learning Center students.

SECONDARY OUTCOMES:
Weight and BMI | 6 and 12 months after intervention
  After students participate in the healthy living program we will measure weight and BMI to evaluate change

CONTACTS AND LOCATIONS:
Overall Officials: Seema Kumar, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials